CLINICAL TRIAL: NCT05358834
Title: Testing Effects of Melatonin on Uterine Contractions in Women
Acronym: MelPreg
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Massachusetts General Hospital (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Elizabeth Klerman MD PhD, Professor, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2021P002926; R01HD107064 (NIH)
Record Dates: First submitted 2022-04-28; First posted 2022-05-03 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Pregnant Women
MeSH Terms: interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Daytime melatonin 0.0 mg (Placebo Comparator): Daytime melatonin 0.0 mg
  Interventions: Dietary Supplement: Placebo
- Daytime melatonin 0.5 mg (Experimental): Daytime melatonin 0.5 mg
  Interventions: Dietary Supplement: Melatonin
- Daytime melatonin 3.0 mg (Experimental): Daytime melatonin 3.0 mg
  Interventions: Dietary Supplement: Melatonin
- Nighttime melatonin 0.0 mg (Placebo Comparator): Nighttime melatonin 0.0 mg
  Interventions: Dietary Supplement: Placebo
- Nighttime melatonin 0.5 mg (Experimental): Nighttime melatonin 0.5 mg
  Interventions: Dietary Supplement: Melatonin

INTERVENTIONS:
Dietary Supplement: Melatonin — Oral melatonin administered as a single pill.
  Arms: Daytime melatonin 0.5 mg; Daytime melatonin 3.0 mg; Nighttime melatonin 0.5 mg
Dietary Supplement: Placebo — Oral placebo administered as a single pill.
  Arms: Daytime melatonin 0.0 mg; Nighttime melatonin 0.0 mg

SUMMARY:
The study will extend recent discoveries that have been made in basic human physiology related to responses melatonin and uterine contractions in late- or full-term pregnant women. The basic physiology work has been conducted in in vitro models of the human myometrium characterizing its responses to melatonin, and in pilot in vivo studies correlating the number of uterine contractions with melatonin concentrations that were manipulated by different types of light exposure. The planned experiments will test a causal link between circulating melatonin levels and uterine contractions in full-term pregnant women by manipulating melatonin levels using exogenous melatonin (i) during the day when endogenous levels of melatonin are very low (Experiment 1), and (ii) during the evening under conditions with lighting that would be expected to suppress the higher evening and nighttime levels of endogenous melatonin (Experiment 2).

ELIGIBILITY:
Inclusion Criteria:

* nulliparity, age between 18 and 35,
* BMI<36 pre-pregnancy,
* ≥38 weeks of pregnancy with a single fetus at time of study.

Exclusion Criteria:

* color blind;
* prescription drugs affecting sleep, melatonin, and/or circadian rhythms (e.g., beta blockers, non-steroidal anti-inflammatory drugs);
* a health or pregnancy related condition that might affect melatonin or uterine contractions;
* medical conditions or medications for which melatonin might be contraindicated or there may be a drug interactions (e.g., Central Nervous System depressants/sedatives, Fluvoxamin (Luvox), medications for diabetes, immunosuppressants, anti-coagulants, Nifedipine, Verapamil).

Note: We cannot list all possible exclusionary criteria. Dr. Carolina Bibbo (co-I), our Obstetrics Investigator at Brigham and Women's Hospital (BWH), will make final determination of suitability including any safety concerns for each potential participant.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Daytime: Total number of uterine contractions | 10 hours
  Daytime: Total number of uterine contractions
Nighttime: Total number of uterine contractions | 4 hours
  Nighttime: Total number of uterine contractions

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth B Klerman, MD PhD, Principal Investigator — MGH
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Per the NIH Policy on Data Sharing, we will make the datasets available to other investigators following publication of the final study results. We will make data available on a public database, such as the NIH-supported National Sleep Research Resource (NSRR; sleepdata.org). Outside investigators should submit their request in writing to the PI. Additional details below in Access Criteria
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Upon request and following publication of the final study results
Access Criteria: Outside investigators should submit their request in writing to the PI. A data-sharing agreement will be required. The request must be in accordance with MGB Policies and Harvard Medical School (HMS) guidelines. Such datasets will not contain identifying information per the regulations outlined in HIPAA, and permission will be obtained from study participants to share their data with researchers outside MGB. Per standard MGB policies, we will require a data-sharing agreement from any investigator or entity requesting the data; this agreement will include: (i) a commitment to using the data only for research purposes and not to identify any individual participant; (ii) a commitment to securing the data using appropriate computer technology; and (iii) a commitment to destroying or returning the data after analyses are completed.